CLINICAL TRIAL: NCT01228669
Title: A Multi-centre, Randomised, Double-blind, Placebo-controlled, Single Dose, Dose Escalation Trial Investigating Safety, Pharmacokinetics and Pharmacodynamics of NNC 0172-0000-2021 Administered Intravenously and Subcutaneously to Healthy Male Subjects and Haemophilia Subjects
Brief Title: Safety of NNC 0172-0000-2021 in Healthy Male Subjects and Subjects With Haemophilia A or B
Acronym: Explorer 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NN7415-3813; 2010-020465-24 (EudraCT Number); U1111-1116-2356 (Other: WHO)
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A; Haemophilia B; Healthy
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: NNC 0172-0000-2021
- B (Experimental)
  Interventions: Drug: NNC 0172-0000-2021
- C (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NNC 0172-0000-2021 — Single dose injected i.v. (into a vein). Each treatment dose is assessed for safety before escalating to next dose
  Arms: A
Drug: NNC 0172-0000-2021 — Single dose injected s.c. (under the skin). Each treatment dose is assessed for safety before escalating to next dose.
  Arms: B
Drug: placebo — Single dose injected i.v. and s.c. Each treatment dose is assessed for safety before escalating to next dose.
  Arms: C

SUMMARY:
This trial is conducted in Europe and Asia. The aim of this clinical trial is to investigate the safety, pharmacokinetics (how the trial drug is distributed in the body) and pharmacodynamics (physiological effects of the drug on the body) of NNC 0172-0000-2021 administered intravenously and subcutaneously to healthy male subjects and subjects with haemophilia A or B

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 50 and 100 kg, both inclusive
* Body mass index (BMI) between 18.0 kg/m2 and 25.0 kg/m2, both inclusive
* For haemophilia subjects only: Diagnosed with severe haemophilia A or B

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product(s) or related products
* Surgery planned to occur during the trial
* Any major and/or orthopaedic surgery within 30 days prior to trial product administration

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-10-25 (Actual); Primary Completion 2012-09-10 (Actual); Study Completion 2012-09-10 (Actual)

PRIMARY OUTCOMES:
Number of adverse Events (AEs), including Serious Adverse Events (SAEs) | from trial product administration until 43 days after trial product administration

SECONDARY OUTCOMES:
Area under the concentration-time curve | from 43 days after trial product administration until 53 days after trial product administration
Adverse Events (AEs), including Serious Adverse Events (SAEs) | from 43 days after trial product administration until 53 days after trial product administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (14):
- Novo Nordisk Investigational Site, Vienna, Austria
- Novo Nordisk Investigational Site, Copenhagen, Denmark
- Germany (2):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Frankfurt/M.
- Novo Nordisk Investigational Site, Milan, Italy
- Novo Nordisk Investigational Site, Kuala Lumpur, Malaysia
- Novo Nordisk Investigational Site, Polokwane, Limpopo, South Africa
- Novo Nordisk Investigational Site, Madrid, Spain
- Novo Nordisk Investigational Site, Malmo, Sweden
- Novo Nordisk Investigational Site, Zurich, Switzerland
- Novo Nordisk Investigational Site, Bangkok, Thailand
- United Kingdom (3):
  - Novo Nordisk Investigational Site, Harrow
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Manchester

REFERENCES:
- [Result] Chowdary P, Lethagen S, Friedrich U, Brand B, Hay C, Abdul Karim F, Klamroth R, Knoebl P, Laffan M, Mahlangu J, Miesbach W, Dalsgaard Nielsen J, Martin-Salces M, Angchaisuksiri P. Safety and pharmacokinetics of anti-TFPI antibody (concizumab) in healthy volunteers and patients with hemophilia: a randomized first human dose trial. J Thromb Haemost. 2015 May;13(5):743-54. doi: 10.1111/jth.12864. Epub 2015 Apr 6. PMID 25641556
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com